CLINICAL TRIAL: NCT00220389
Title: Two Phase Extension Trial of SP668 to Investigate the Safety and Tolerability of Sustained Release Fesoterodine in Subjects With Overactive Bladder(OAB): a Double-Blind Phase Followed by an Open-Label Extension Phase
Brief Title: Two Phase Extension Trial of SP668 to Investigate the Safety and Tolerability of Sustained Release Fesoterodine in Subjects With Overactive Bladder: a Double-Blind Phase Followed by an Open-Label Extension Phase
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: SP669
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Last update posted 2008-10-16 (Estimated); Status verified 2008-10

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive

INTERVENTIONS:
Drug: SPM 907

SUMMARY:
This extension trial of SP668 consists of two phases: double-blind treatment and open-label extension. The trial provides subjects the option of long-term treatment with sustained release (SR) fesoterodine (SPM 907) and to assess long-term subject safety, tolerability and efficacy.

Double-Blind: Subjects remained on either fesoterodine 4mg, 8mg or 12mg depending on their dose assignment in SP668. Previous SP668 placebo subjects received fesoterodine 4mg.

Open-Label: Subjects received fesoterodine 8mg with a one time option to reduce the dose to 4mg and a one time option to increase again to 8mg.

The primary variables focus on long-term safety and tolerability and include the observation and assessment of adverse events, residual urinary volumes, laboratory parameters, changes in ECG, physical and urological examinations and subject's assessment of treatment tolerance.

Secondary efficacy variables include various parameters derived from micturition diaries, count of subjects and their dose choice throughout the trial and subject's assessment of treatment efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Overactive bladder

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2003-06; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brooke Derby, Study Director — UCB Pharma
Locations (1):
- Schwarz, RTP, North Carolina, United States